CLINICAL TRIAL: NCT02383680
Title: Yellow Fever Vaccination Under Low Dose Methotrexate Therapy - a Multi-Center Prospective Observational Controlled Pilot Study
Brief Title: Yellow Fever Vaccination Under Low Dose Methotrexate Therapy
Acronym: MTX_YF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Swiss Tropical & Public Health Institute (Other); Kantonsspital Aarau (Other); Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Geneva (Other); Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor
Other Study IDs: CS_2014_01
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatic; Dermatologic Disorders
Keywords: Methotrexate therapy
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients under low dose methotrexate therapy: Patients with various underlying conditions (e.g. rheumatic diseases, dermatologic diseases) who have an indication for yellow fever vaccination
  Interventions: Biological: Yellow Fever Vaccination
- Healthy controls: Healthy travelers who have an indication for yellow fever vaccination
  Interventions: Biological: Yellow Fever Vaccination

INTERVENTIONS:
Biological: Yellow Fever Vaccination — The Yellow Fever vaccination is actually not part of the study. Only individuals who have an indication for yellow fever vaccination according to Swiss vaccination recommendations will be enrolled. Study procedures will include blood collection to measure antibody development and viremia as well as data collection on possible side effects.

SUMMARY:
Travelers (n = 30, 15 taking low-dose methotrexate (MTX), 15 healthy controls (HC), seeking travel advice in one of the following Swiss Travel Centers (Aarau, Basel, Bern, Geneva, Lausanne, Zurich) and who have an indication for yellow fever (YF) vaccination according to the Swiss Federal Office of Public Health's vaccination recommendations are invited to participate in this study. After signing the consent form (i) YF viremia and (ii) anti-YF antibody production in patients taking low-dose MTX and HC will be compared after YF vaccination. It will be analyzed whether the percentage of people with protective antibodies differs between the two groups and (iii) vaccine side effects will be compared between the groups.

DETAILED DESCRIPTION:
The study will be conducted in the form of a multi-center open-label prospective observational controlled pilot study. 15 patients under low dose methotrexate treatment and 15 healthy controls with an indication for yellow fever vaccination will be included. The study duration will be 28 days for each subject and will consist of 6 clinical visits on days 0, 3, 7, 10, 14 and 28.

YF antibodies will be measured on days 0, 7, 10, 14 and 28; viremia will be measured on days 3, 7, 10, 14 and 28.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Indication for yellow fever vaccination according to Swiss FOPH recommendations
* Individuals under low dose MTX (≤20mg/week) therapy or healthy individuals
* Male and Female travelers ≥18 years to <60 years of age

Exclusion Criteria:

* Contraindications on ethical grounds
* Women who are pregnant or breast feeding
* Contraindication against yellow fever vaccination (e.g. hypersensitivity against vaccine ingredient)
* Current treatment with other immunosuppressive agent apart from low dose methotrexate
* Alemtuzumab or rituximab in the last year
* TNF-blocking therapy in past three months
* Immunocompromising condition in healthy control
* Other immunocompromising condition than MTX treatment itself and the underlying disease in patients under MTX
* Previous yellow fever vaccination
* No indication for yellow fever vaccination according to Swiss travel vaccination recommendations
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Travelers seeking pre-travel advice with an indication for yellow fever vaccination will be addressed in 6 Swiss Travel Clinics of the Cantonal Hospital Aarau, the University Hospital in Bern, the University of Zurich, teh University Hospital of Geneva and the Swiss Tropical and Public Health Instutute in Basel
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Quantitative viremia in blood in travelers under low dose methotrexate (≤20mg/week) and healthy travelers | days 3, 7, 10 and 14 and 28
  Serum samples will be collected for PCR
Quantitative yellow fever specific neutralizing antibodies in blood of travelers under low dose methotrexate therapy (≤20mg/week) and healthy travelers | days 0, 7, 10, 14 and 28
  Serum samples will be collected for measurement of neutralizing antibodies

SECONDARY OUTCOMES:
Determination of the percentage of travelers with an antibody level of >0.7 LNI (>0.5 IU/ml) in both groups | days 0, 7, 10, 14, 28
Assessment of safety by determining the severity and quantity of adverse vaccine reactions such as local and systemic reactions in both study groups | Throughout day 28 after vaccination
  Local and systemic vaccine reactions will be collected in a diray card filled out by the participant

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hatz, Prof MD, Principal Investigator — University of Zurich, Epidemiolgy, Biostatistics and Prevention Institute
Locations (6):
- Switzerland (6):
  - Kantonsspital Aarau, Aarau, Canton of Aargau
  - Swiss Tropical and Public Health Institute, Basel, Canton of Basel-City
  - Universitätsklinik für Infektiologie Inselspital, Bern, Canton of Bern
  - Médecine Tropicale et Humanitaire Hôpitaux Universitaires de Genève, Geneva, Canton of Geneva
  - University of Zurich, Epidemiology, Biostatistics and Prevention Institute, Zurich, Canton of Zurich
  - PMU | Policlinique médicale universitaire CHUV | Service des maladies infectieuses, Département de médecine, Lausanne